CLINICAL TRIAL: NCT04442464
Title: Intraocular Pressure in Ocular Hypertensives With Scleral Lens Wear
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cherie B. Nau, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-004974
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study Eye (Experimental): One eye will be randomly selected to wear the scleral lenses to be worn during study measurements
  Interventions: Device: Scleral Lens
- Control Eye (No Intervention): Non-lens wearing eye

INTERVENTIONS:
Device: Scleral Lens — 15.0 mm diagnostic spherical rigid contact lens
  Arms: Study Eye

SUMMARY:
The purpose of this study is to determine if short-term wear of a spherical rigid contact lens, called a scleral lens, will raise intraocular pressure in ocular hypertensive patients.

DETAILED DESCRIPTION:
This is a randomized, self-controlled study designed to compare effectiveness of a scleral lens on intraocular pressure. In this study, all participants have one eye randomly selected to wear the scleral lenses during study measurements and the other eye serves as the control, non-lens wearing eye.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension (IOP >22 in each eye during at least two visits over the previous 3 years)
* May have had cataract extraction and intraocular lens (IOL)
* Not on topical medication for glaucoma
* No History of ALT/SLT
* Any Age, 18 years or older
* History of contact lens wear (except scleral lenses), as long as they are willing to not wear their lenses the day of the study

Exclusion Criteria:

* On topical medication for glaucoma
* Eye disease
* Inability to wear scleral lenses
* Any intraocular surgery other than uncomplicated cataract extraction.
* Known allergy to proparacaine eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Nau, OD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eye
Period: Overall Study
Arm/Group | Study Eye | Control Eye
Started | 1; 1 Eye | 1; 1 Eye
Completed | 1; 1 Eye | 1; 1 Eye
Not Completed | 0; 0 Eye | 0; 0 Eye

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants had one eye randomly selected to wear the scleral lenses during study measurements and the other eye served as the control, non-lens wearing eye.
  Scleral Lens: 15.0 mm diagnostic spherical rigid contact lens
Arm/Group | All Study Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Intraocular pressure measured in millimeters of mercury (mm Hg)
Time Frame: 4 hours
Measure: Number; unit: mmHg
Units Other Than Participants: Eye
Arm/Group | Study Eye | Control Eye
Number analyzed (Participants) | 1 | 1
Number analyzed (Eye) | 1 | 1
mmHg
  Baseline | 24.0 | 23.5
  4 hours | 21.2 | 21.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 1 day on all participants.
Arm/Group | Study Eye | Control Eye
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study terminated due to lack of recruitment and only one participant was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT04442464/Prot_SAP_000.pdf